CLINICAL TRIAL: NCT02819557
Title: A Phase 2 Study of the Safety, Pharmacokinetics, and Pharmacodynamics of Ataluren (PTC124®) in Patients Aged ≥2 to <5 Years Old With Nonsense Mutation Dystrophinopathy
Brief Title: Study of Ataluren in ≥2 to <5 Year-Old Male Participants With Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-030-DMD
Record Dates: First submitted 2016-06-16; First posted 2016-06-30 (Estimated); Results first posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ataluren (Experimental): Participants will be administered ataluren orally at a dose of 10 milligrams/kilograms (mg/kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening (for a total of 40 mg/kg/day) for up to 52 weeks. Dose will be provided based upon the weight of each participant, which will be assessed every 12 weeks.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — White to off-white powder for oral suspension.
  Other Names: PTC124; Translarna

SUMMARY:
This is a Phase 2, multiple-dose, open-label study evaluating the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of ataluren in participants aged ≥2 to <5 years old with Duchenne muscular dystrophy (DMD) caused by a nonsense mutation in the dystrophin gene.

DETAILED DESCRIPTION:
In nonsense mutation DMD (nmDMD), early start of treatment is important and necessary and, therefore, it is relevant to understand the correct and tolerable dose in this age group, particularly since ataluren is dosed by weight. This study included a 4-week screening period, a 52-week treatment period (the first 4 weeks of which included PK parameters), and a 4-week follow-up period for participants who completed the treatment period (60 weeks total duration). The objective of the extension period (treatment period after PK parameters have been completed) was to assess the long-term safety of chronic administration of ataluren in this participant population.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥2 to <5 years of age
* Body weight ≥12 kg
* Diagnosis of DMD
* Nonsense mutation in at least 1 allele of the dystrophin gene

Exclusion Criteria:

* Participation in any other drug or device clinical investigation
* Ongoing use of prohibited concomitant medications

Ages: 2 Years to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bibbiani, MD, Study Director — PTC Therapeutics
Locations (6):
- United States (6):
  - Child Neuro NWF, Gulf Breeze, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Medical Center Dallas, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged ≥2 to <5 years old with Duchenne muscular dystrophy (DMD) caused by a nonsense mutation in the dystrophin gene were recruited for this study.
Pre-assignment Details: Participants in the Evaluable Population included all participants who received at least 1 dose of ataluren and had a baseline and at least 1 postbaseline measurement for Timed Function Test (TFT), North Star Ambulatory Assessment (NSAA), or response to the palatability of ataluren questions.
Groups:
- Ataluren: Participants were administered ataluren orally at a dose of 10 milligrams/kilograms (mg/kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening (for a total of 40 mg/kg/day) for up to 52 weeks. Dose was provided based upon the weight of each participant, which was assessed every 12 weeks.
Period: Overall Study
Arm/Group | Ataluren
Started | 14
Safety Population (All participants who received at least 1 dose of ataluren.) | 14
Pharmacokinetics (PK) Population (All participants who received at least 1 dose of ataluren and had at least 1 PK concentration value.) | 14
Evaluable Population (Received ≥1 dose, baseline and a postbaseline TFT, NSAA, or answer to ataluren palatability question) | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of ataluren (Safety Population).
Groups:
- Ataluren: Participants were administered ataluren orally at a dose of 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening (for a total of 40 mg/kg/day) for up to 52 weeks. Dose was provided based upon the weight of each participant, which was assessed every 12 weeks.
Arm/Group | Ataluren
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.4 (0.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), TEAEs Leading to Discontinuation, and Serious Adverse Events (SAEs)
Description: A TEAE was any untoward medical occurrence or undesirable event that begins or worsens following administration of study drug, whether or not considered related to study drug by Investigator. An SAE was an adverse event (AE) resulting in any of the following outcomes or deemed significant for any other reason, death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying) or persistent or significant disability/incapacity not related to dystrophinopathy. An event was not reported as an SAE, if event was exclusively a relapse or expected change or progression of baseline dystrophinopathy. AEs included both SAEs and nonserious AEs. AEs classified according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 and coded using Medical Dictionary for Regulatory Activities. A summary of SAEs and all non-serious AEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline up to Week 56
Population: All participants who received at least 1 dose of ataluren (Safety Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 14
Participants
  At least 1 TEAE | 14
  Mild TEAE | 5
  Moderate TEAE | 8
  Severe TEAE | 1
  TEAE Related to Study Drug | 5
  TEAE Leading to Participant Study Discontinuation | 0
  Serious TEAE | 0

2. Primary Outcome: Number of Participants With a Clinically Meaningful Abnormal Clinical Laboratory (Biochemistry, Hematology, and Urinalysis) Parameter
Description: Clinical laboratory results that were considered clinically meaningful were to be determined by the Investigator and Sponsor. Biochemistry parameters included sodium, potassium, chloride, bicarbonate, blood urea nitrogen, creatinine, magnesium, calcium, phosphorus, uric acid, glucose, total protein, albumin, bilirubin (total, direct, and indirect), aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transferase, creatine kinase, lactate dehydrogenase, alkaline phosphatase, total cholesterol, high-density lipoprotein, low-density lipoprotein, triglycerides, and cystatin C. Hematology parameters included white blood cell count with differential, hemoglobin, hematocrit, other red cell parameters, and platelet count. Urinalysis parameters included pH, specific gravity, glucose, ketones, blood, protein, urobilinogen, bilirubin, nitrite, and leukocyte esterase. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 56
Population: All participants who received at least 1 dose of ataluren (Safety Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 14
Participants | 0

3. Primary Outcome: Number of Participants With a Clinically Meaningful Abnormal Electrocardiogram (ECG) Test Results
Description: ECG results that were considered clinically meaningful were to be determined by the Investigator. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 56
Population: All participants who received at least 1 dose of ataluren (Safety Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 14
Participants | 0

4. Primary Outcome: Number of Participants With a Dose-Limiting Toxicity as Measured by Hepatic and Renal Toxicity
Description: Dose-limiting toxicity was measured through clinical evaluations for potential hepatic and renal toxicities. The clinical evaluations included the following:
  * Hepatic: The participant's medical history, hepatitis screening results, all clinical blood values (particularly serum bilirubin, gamma-glutamyl transferase [GGT], aspartate aminotransferase [AST], and alanine aminotransferase [ALT] values), and all concomitant medications were reviewed.
  * Renal: The participant's medical history, all clinical blood and urine renal values, serum electrolytes, medications, and potential pre- or post-renal conditions were reviewed.
Time Frame: Baseline up to Week 56
Population: All participants who received at least 1 dose of ataluren (Safety Population).
Measure: Number; unit: participants
Arm/Group | Ataluren
Number analyzed (Participants) | 14
participants | 0

5. Secondary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration From Time Zero up to 6 Hours After the Morning Dose (Cmax0-6hr)
Description: Ataluren concentrations in plasma were analyzed using a validated high performance liquid chromatography-tandem mass spectrometry (HPLC-MS/MS) method.
Time Frame: 0 (predose), 1, 2, 4, and 6 (postdose) hours on Days 1 and 28
Population: All participants who received at least 1 dose of ataluren and had at least 1 PK concentration datum (PK Population).
Measure: Mean (Standard Deviation); unit: microgram/milliliter (µg/mL)
Arm/Group | Ataluren
Number analyzed (Participants) | 14
microgram/milliliter (µg/mL)
  Day 1 | 15.95 (9.51)
  Day 28 | 12.54 (4.43)

6. Secondary Outcome: Pharmacokinetics: Time to Reach Maximum Observed Plasma Concentration From Time Zero up to 6 Hours After the Morning Dose (Tmax0-6hr)
Description: Ataluren concentrations in plasma were analyzed using a validated HPLC-MS/MS method.
Time Frame: 0 (predose), 1, 2, 4, and 6 (postdose) hours on Days 1 and 28
Population: All participants who received at least 1 dose of ataluren and had at least 1 PK concentration datum (PK Population).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ataluren
Number analyzed (Participants) | 14
hours
  Day 1 | 3.84 (1.82)
  Day 28 | 2.72 (1.98)

7. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero up to 10 Hours After the Morning Dose (AUC0-10hr)
Description: Ataluren concentrations in plasma were analyzed using a validated HPLC-MS/MS method. AUC0-10hr was measured using the linear trapezoidal rule during the ascending portion of the curve and the log-trapezoidal rule during the descending portion of the curve.
Time Frame: 0 (predose), 1, 2, 4, 6, 8, and 10 (postdose) hours on Days 1 and 28
Population: All participants who received at least 1 dose of ataluren and had at least 1 PK concentration datum (PK Population).
Measure: Mean (Standard Deviation); unit: hour*μg/mL
Arm/Group | Ataluren
Number analyzed (Participants) | 14
hour*μg/mL
  Day 1 | 101.64 (58.52)
  Day 28 | 82.13 (27.43)

8. Secondary Outcome: Pharmacokinetics: Concentration at the End of the First (Morning) Dose Interval (Ctrough6hr)
Description: Ataluren concentrations in plasma were analyzed using a validated HPLC-MS/MS method.
Time Frame: 0 (predose), 1, 2, 4, and 6 (postdose) hours on Days 1 and 28
Population: All participants who received at least 1 dose of ataluren and had at least 1 PK concentration datum (PK Population).
Measure: Mean (Standard Deviation); unit: microgram per milliliter (µg/ml)
Arm/Group | Ataluren
Number analyzed (Participants) | 14
microgram per milliliter (µg/ml)
  Day 1 | 9.12 (8.88)
  Day 28 | 5.43 (3.15)

9. Secondary Outcome: Change From Baseline in Proximal Muscle Function as Assessed by Speed During TFTs
Description: TFTs included time to stand from supine position (rise to standing), time to run/walk 10 meters (m), and time to ascend/descend 4 stairs. A decrease from baseline reflects faster completion of the functional task and, thus, better muscle function. If the time taken to perform a test exceeded 30 seconds or if a participant could not perform the test due to disease progression (PD), a value of 30 seconds was used.
Time Frame: Baseline, Week 28 and Week 52
Population: All participants who received at least 1 dose of ataluren and had a baseline and at least 1 postbaseline measurement for TFT, NSAA, or response to the palatability of ataluren questions (Evaluable Population) and had evaluable data for the applicable timed function test.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ataluren
Number analyzed (Participants) | 14
seconds
  Rise to Standing, Baseline | 7.2 (7.21)
  Rise to Standing, Change from Baseline at Week 28: number analyzed (Participants) | 13
  Rise to Standing, Change from Baseline at Week 28 | -3.1 (6.47)
  Rise to Standing, Change from Baseline at Week 52 | -3.1 (6.50)
  Walk/Run 10 m, Baseline | 6.6 (2.37)
  Walk/Run 10 m, Change from Baseline at Week 28: number analyzed (Participants) | 13
  Walk/Run 10 m, Change from Baseline at Week 28 | -0.8 (1.54)
  Walk/Run 10 m, Change from Baseline at Week 52 | -1.1 (1.35)
  Ascend 4 Stairs, Baseline | 7.1 (6.95)
  Ascend 4 Stairs, Change from Baseline at Week 28: number analyzed (Participants) | 13
  Ascend 4 Stairs, Change from Baseline at Week 28 | -1.8 (4.85)
  Ascend 4 Stairs, Change from Baseline at Week 52 | -2.6 (5.00)
  Descend 4 Stairs, Baseline: number analyzed (Participants) | 13
  Descend 4 Stairs, Baseline | 7.5 (3.95)
  Descend 4 Stairs, Change from Baseline at Week 28: number analyzed (Participants) | 12
  Descend 4 Stairs, Change from Baseline at Week 28 | -0.6 (1.93)
  Descend 4 Stairs, Change from Baseline at Week 52: number analyzed (Participants) | 13
  Descend 4 Stairs, Change from Baseline at Week 52 | -2.2 (2.58)

10. Secondary Outcome: Change From Baseline in Physical Function as Measured by the NSAA
Description: NSAA consists of 17 activities, including items assessing abilities necessary to remain functionally ambulant (that is, ability to rise from floor, to get from lying to sitting/sitting to standing, and that are known to progressively deteriorate); items that can be partly present in DMD early stages (that is, assessing head raise and standing on heels); and a number of activities such as hopping, jumping, and running. Since the boys were <5 years old, revised 16 point, 8-point, and 3-point scales were used over the 17 point scale. Scores for evaluations=0 (Unable to achieve independently), 1 (Modified method but achieved goal independent of physical assistance), or 2 (Normal, no obvious modification of activity). Maximum total score for the 16-point scale=32, 8-point scale=16, and 3-point scale=6. If an activity couldn't be performed due to PD/loss of ambulation, a score of 0 was assigned. Change from Baseline calculated by subtracting Baseline value from value at Week 28 and Week 52.
Time Frame: Baseline, Week 28 and Week 52
Population: All participants who received at least 1 dose of ataluren and had a baseline and at least 1 postbaseline measurement for TFT, NSAA, or response to the palatability of ataluren questions (Evaluable Population) and had evaluable NSAA data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 14
units on a scale
  16-Point Scale, Baseline | 16.0 (4.66)
  16-Point Scale, Change from Baseline at Week 28: number analyzed (Participants) | 13
  16-Point Scale, Change from Baseline at Week 28 | 3.5 (3.43)
  16-Point Scale, Change from Baseline at Week 52 | 5.5 (4.43)
  8-Point Scale, Baseline | 10.5 (2.56)
  8-Point Scale, Change from Baseline at Week 28: number analyzed (Participants) | 13
  8-Point Scale, Change from Baseline at Week 28 | 1.5 (1.39)
  8-Point Scale, Change from Baseline at Week 52 | 2.3 (2.13)
  3-Point Scale, Baseline | 5.4 (0.63)
  3-Point Scale, Change from Baseline at Week 28: number analyzed (Participants) | 13
  3-Point Scale, Change from Baseline at Week 28 | 0.5 (0.78)
  3-Point Scale, Change from Baseline at Week 52 | 0.3 (0.73)

11. Secondary Outcome: Change From Baseline in Height of Participants at Weeks 4, 16, 28, 40, 52, and 56
Time Frame: Baseline, Weeks 4, 16, 28, 40, 52, and 56
Population: All participants who received at least 1 dose of ataluren (Safety Population) and had evaluable height data.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Ataluren
Number analyzed (Participants) | 14
centimeters
  Baseline | 99.43 (5.278)
  Change at Week 4 | 0.83 (1.595)
  Change at Week 16 | 1.84 (1.466)
  Change at Week 28 | 3.11 (1.386)
  Change at Week 40: number analyzed (Participants) | 13
  Change at Week 40 | 3.82 (1.506)
  Change at Week 52 | 5.95 (2.096)
  Change at Week 56 | 6.04 (2.075)

12. Secondary Outcome: Change From Baseline in Weight of Participants at Weeks 4, 16, 28, 40, 52, and 56
Time Frame: Baseline, Weeks 4, 16, 28, 40, 52, and 56
Population: All participants who received at least 1 dose of ataluren (Safety Population) and had evaluable weight data.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ataluren
Number analyzed (Participants) | 14
kg
  Baseline | 16.99 (3.257)
  Change at Week 4 | -0.04 (0.502)
  Change at Week 16 | 0.73 (0.974)
  Change at Week 28 | 1.16 (0.940)
  Change at Week 40: number analyzed (Participants) | 13
  Change at Week 40 | 1.39 (0.882)
  Change at Week 52 | 1.90 (1.259)
  Change at Week 56 | 2.13 (1.340)

13. Secondary Outcome: Change From Baseline in Body Mass Index of Participants at Weeks 4, 16, 28, 40, 52, and 56
Description: Body mass index is an estimate of body fat based on body weight divided by height squared.
Time Frame: Baseline, Weeks 4, 16, 28, 40, 52, and 56
Population: All participants who received at least 1 dose of ataluren (Safety Population).
Measure: Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)
Arm/Group | Ataluren
Number analyzed (Participants) | 14
kilograms per square meter (kg/m^2)
  Baseline | 17.094 (2.2196)
  Change at Week 4 | -0.346 (0.6804)
  Change at Week 16 | 0.026 (0.3822)
  Change at Week 28 | 0.030 (0.5567)
  Change at Week 40: number analyzed (Participants) | 13
  Change at Week 40 | 0.008 (0.6399)
  Change at Week 52 | -0.186 (0.9237)
  Change at Week 56 | 0.015 (1.2161)

14. Secondary Outcome: Ataluren Palatability Characteristics as Determined by a Parent/Caregiver Questionnaire
Description: To assess palatability characteristics, participants/parents or guardians were asked to provide a response of "Strongly disagree", "Disagree", "Neither agree or disagree", "Agree", or "Strongly Agree" to the following 3 questions:
  Question 1. "Is the medicine palatable?"
  Question 2. "On the basis of reaction / facial expression of your child, do you think that the medication is pleasant?"
  Question 3."You sometimes have problems in giving the medication to your child because he/she refuses to take it or throws it up?"
Time Frame: Baseline up to Week 28
Population: All participants who received at least 1 dose of ataluren and had a baseline and at least 1 postbaseline measurement for TFT, NSAA, or response to the palatability of ataluren questions (Evaluable Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 14
Participants
  Question 1, Strongly disagree | 0
  Question 1, Disagree | 0
  Question 1, Neither Agree nor Disagree | 2
  Question 1, Agree | 0
  Question 1, Strongly agree | 0
  Question 1, No Response | 12
  Question 2, Strongly disagree | 0
  Question 2, Disagree | 2
  Question 2, Neither Agree nor Disagree | 2
  Question 2, Agree | 6
  Question 2, Strongly Agree | 4
  Question 2, No response | 0
  Question 3, Strongly Disagree | 5
  Question 3, Disagree | 7
  Question 3, Neither agree or disagree | 0
  Question 3, Agree | 2
  Question 3, Strongly Agree | 0
  Question 3, No response | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 56
Description: Adverse events were collected from all participants who received at least 1 dose of ataluren (Safety Population).
Arm/Group | Ataluren
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 14/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=14)
Abdominal Pain Upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 1
Gait Disturbance (General disorders) | 1
Pyrexia (General disorders) | 6
Bronchitis Viral (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Croup Infectious (Infections and infestations) | 1
Ear Infection (Infections and infestations) | 5
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis Norovirus (Infections and infestations) | 1
Gingival Abscess (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 4
Pharyngitis Streptococcal (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2
Viral Rash (Infections and infestations) | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1
Hepatic Enzyme Increased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Abnormal Behaviour (Psychiatric disorders) | 1
Enuresis (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Rash Generalised (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the Sponsor for review. The Sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-01-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT02819557/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT02819557/SAP_001.pdf